CLINICAL TRIAL: NCT03696277
Title: A Phase II Trial of Stereotactic Ablative Radiation Therapy (SAbR) for Patients With Oligo-progressive Renal Cell Cancer (RCC).
Brief Title: SAbR For Oligo-Progressive Renal Cell Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052018-001
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Oligoprogressive Renal Cell Carcinoma
Keywords: Stereotactic, Radiotherapy,

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic ablative body radiation (SABR) (Experimental): SAbR will be used to treat all sites of measurable metastases. New sites of metastasis will be treated if deemed appropriate by both medical and radiation oncologists with SAbR.
  Interventions: Radiation: Stereotactic ablative body radiation (SABR)

INTERVENTIONS:
Radiation: Stereotactic ablative body radiation (SABR) — SAbR treatment regimens including ≥25Gy x1 fraction, ≥12Gy x 3 fractions, or ≥8Gy x 5 fractions.

SUMMARY:
Metastatic kidney cancer patients on systemic therapy often develop resistance to limited sites that leads to changing of the systemic therapy. Local therapy to the sites of progression may allow patients to continue on the same systemic therapy that is otherwise effective and being tolerated well.

Hypothesis:

Stereotactic ablative radiation (SAbR) can delay the change of systemic therapy with oligoprogressive renal cell cancer (RCC) and improve progression free survival (PFS).

Primary Objectives:

• To evaluate the benefit of SAbR for oligo-progressive mRCC (Metastatic Renal Cell Cancer).

Secondary Objectives:

• To measure the toxicity, safety and tolerance of concurrent systemic therapy and SAbR for mRCC patients and its impact on quality of life.

DETAILED DESCRIPTION:
The study is a prospective phase II, single arm, open label trial evaluating Stereotactic Ablative Radiation Therapy (SAbR) for patients with oligo-progressive RCC (Renal Cell Cancer).

Problem Statements:

* Can local therapy (SAbR) for oligoprogression delay the change of systemic therapy if progression is minimal to the progressive sites?
* Safely delaying the change of systemic therapy can have significant quality of life benefits for patients with oligo-progressive RCC.
* Can SAbR potentially improve progression free survival in oligoprogressive RCC patients?

Primary Endpoint:

• Time to change of systemic therapy.

Secondary Endpoint:

* PFS on subsequent systemic therapy (PFS-SST) after progression on SAbR.
* Overall survival(OS).
* Toxicity, safety and tolerance.
* Impact on health-related quality of life (HRQoL).

Sample Size: 20 Patients

Statistical Analysis: Time to event will be estimated using the Kaplan-Meier approach along with the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology proven renal cell carcinoma and radiographic confirmation of metastatic renal cell carcinoma
2. Patients must have drug responsive RCC as determined by treating medical or radiation oncologist after at least one set of scans.
3. Must be on systemic therapy with radiographic scans to verify olio-progression of ≤3 sites and ≤ 30% of all sites.

   • Any FDA approved systemic therapy for RCC is allowed. Currently these include small molecule tyrosine kinase inhibitors (TKIs) targeting the vascular endothelial growth factor (VEGF) pathway (sunitinib, pazopanib, cabozantinib, axitinib, sorafenib), monoclonal antibody targeting the same pathway (bevacizumab), the mammalian target of rapamycin pathway (temsirolimus, everolimus), Immune checkpoint inhibitors (Nivolumab and Nivolumab concurrent with Ipilimumab, Lenvatinib in combination with everolimus and nivolumab).
4. Must be at least 18 years old
5. ECOG 0-2; or KPS > 60
6. Currently receiving 1st - 4th line of systemic therapy

   • Any of the above listed systemic therapy is allowed as long as they are being used in the 1st-4th line setting.
7. Ability to understand and the willingness to sign a written informed consent.
8. Acceptable tolerability of ongoing therapy as decided by the treating medical oncologist
9. Patient must have a desire to continue ongoing therapy
10. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    * A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

      * Has not undergone a hysterectomy or bilateral oophorectomy; or
      * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months

Exclusion Criteria:

* Subjects with ≥3 unfavorable prognostic factors defined by IMDC (International Metastatic Renal Cell Carcinoma).
* Subjects with history of or new brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Time to change of systemic therapy | 2 Years
  SAbR for oligo-progression will be measured to delay the change of systemic therapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 years
  Progression-Free Survival on systemic therapy started (PFS-ST) after progression on SAbR with existing or new progression at >3 or >30% of all lesions.
Overall survival | 6 Years
  Overall Survival (OS), which is defined as the time between date of registration and the date of death due to any cause.
Number of participants with adverse events | 6 Years
  Severity or Toxicity will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0. The consequences of toxicity should all be graded 1-5 according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Health-related quality of life (HRQOL) | 6 Years
  HRQoL will be measured using Functional Assessment of Cancer Therapy (FACT-G)questionnaire. The FACT-G is a 28-item questionnaire that uses 5-point Likert-type response choices (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Possible scores range from 0-4, where higher scores indicate better outcome.
Health-related quality of life (HRQOL) | 6 years
  HRQoL is measured using EuroQoL- 5 Dimension (EQ-5D) questionnaire. EQ-5D is a patient self-administrated questionnaire. The first part consists of 5 items covering 5 dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be graded on 3 levels: 1-no problems, 2-moderate problems, and 3-extreme problems. Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 health states to which unconsciousness and death are added. The 5-item index score is transformed into a utility score between. Possible scores range from 0-1, where higher score indicates better outcomes ( 0 ="Worst health state," and 1="Best health state." )
Quality of life (QOL) | 6 years
  HRQoL will be measured using Kidney Symptom Index (FKSI) questionnaire. FKSI is a 15 question validated symptom index for kidney cancer patients that uses 5-point Likert-type response choices (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Possible scores range from 0-4, where higher scores indicate better outcome.
Quality of life with cost involved | 6 years
  QOL will be measured using Cost & Convenience Questionnaire. This outcome measure will not be used and data will not be collected or analyzed because of a protocol amendment Version 4 approved on 06/26/2020.
Local control | 6 years
  Radiographic progression with >20% increase in the longest diameter of the treated lesions.
  This outcome measure will not be used and data will not be collected or analyzed because this outcome measure was added in error at the time of the initial registration.

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States